CLINICAL TRIAL: NCT02654873
Title: Is Routine Use of Histopathological Examination Necessary After Cholecystectomy ?
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Collaborators: Bezmialem Vakif University (Other); Istanbul Training and Research Hospital (Other Government); Erzincan University (Other); Arnavutkoy State Hospital (Other); Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, M.D., Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: Sislietfal
Record Dates: First submitted 2016-01-10; First posted 2016-01-13 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Cholelithiasis
Keywords: histopathology; gallbladder; specimen
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cholecystectomy specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Benign: Benign pathology specimens with macroscopically
- Suspicious: Suspicious group includes the conditions such as increasing of the gallbladder wall thickness, having calcifications or polyps in the gallbladder.
- Malign: Malign group includes the conditions such as detecting mass or irregularities in the gallbladder wall.

SUMMARY:
Cholecystectomy has been made with benign conditions usually. The aim of this study is to compare the macroscopic evaluations of the cholecystectomy specimens with it's histopathological examinations.

DETAILED DESCRIPTION:
Cholecystectomy is one of the most frequently performed surgery in the world and often made with benign conditions. Routinely cholecystectomy specimens sent for histopathologic examination. The histopathologic examination of the cholecystectomy specimens are benign in most of the cases and the incidental malignancy of the gallbladder is 2-2.9% in the literature. The histopathologic evaluations of the gallbladder come with additional workload for pathology and surgery departments. Also there is additional cost for the patients. Because of that the idea of selective histopathologic examination has been raised.

ELIGIBILITY:
Inclusion Criteria:

* Subject has cholelithiasis

Exclusion Criteria:

* Subject has acute cholecystitis
* Subject has perforated gallbladder
* Subject has malignancy
* Subject has polyps in the gallbladder
* Subject has increasing wall thickness of the gallbladder
* Subject has malignancy in the preoperative ultrasonography in the gallbladder
* Subject has pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 patients who is operated with non inflamated cholelithiasis will be included to this study.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-12; Primary Completion 2017-10 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The comparison of macroscopic and histopathologic examination of the cholecystectomy specimen with 1000 cases | 15 days
  The 1000 cholecystectomy specimens will be evaluated macroscopically by two experienced surgeons with a longitudinal incision to the gallbladder. The specimens will be grouped as benign, suspicious, malign according to the surgeon's decision. To confirm the surgeon's macroscopic evaluation, all of the specimens will be evaluated histopathologically. The results of macroscopic and histopathological examinations will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, M.D., Study Director — Sisli Etfal Training and Research Hospital; Huseyin Bektasoglu, M.D., Principal Investigator — Bezmialem Vakif University
Locations (6):
- Turkey (Türkiye) (6):
  - Bursa Yuksek Ihtisas Training and Research Hospital, Bursa
  - Erzincan University, Erzincan
  - Bezmialem Vakif University, Istanbul
  - Sisli Etfal Training and Research Hospital, Istanbul
  - Arnavutkoy State Hospital, Istanbul
  - Istanbul Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
Because the time period of this study is very short

REFERENCES:
- [Background] Elshaer M, Gravante G, Yang Y, Hudson S, Thomas K, Sorge R, Al-Hamali S, Kelkar A, Ebdewi H. Routine versus selective histologic analysis of gallbladder specimens for the detection of incidental gallbladder cancers. A retrospective review over 9 years of activity with a special focus on patients' age. Am J Surg. 2014 Sep;208(3):444-9. doi: 10.1016/j.amjsurg.2013.12.038. Epub 2014 Apr 3. PMID 24811928
- [Background] Siddiqui FG, Memon AA, Abro AH, Sasoli NA, Ahmad L. Routine histopathology of gallbladder after elective cholecystectomy for gallstones: waste of resources or a justified act? BMC Surg. 2013 Jul 8;13:26. doi: 10.1186/1471-2482-13-26. PMID 23834815
- [Result] Deng YL, Xiong XZ, Zhou Y, Shrestha A, Li FY, Cheng NS. Selective histology of cholecystectomy specimens--is it justified? J Surg Res. 2015 Jan;193(1):196-201. doi: 10.1016/j.jss.2014.07.039. Epub 2014 Jul 24. PMID 25151466